CLINICAL TRIAL: NCT03106324
Title: A Prospective Non-interventional Post-authorization Safety Study (PASS) of Lenalidomide in Previously Untreated Adult Multiple Myeloma Patients Who Are Not Eligible for Transplant ("Transplant Noneligible" [TNE])
Brief Title: A Safety Study of Lenalidomide in Previously Untreated Adult Multiple Myeloma Patients Who Are Not Eligible for Transplant
Status: Active, not recruiting | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-5013-MM-034; U1111-1194-5810 (Other: World Health Organization)
Record Dates: First submitted 2017-03-29; First posted 2017-04-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Non transplant eligible; Revlimid; PASS; Non-interventional; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TNE NDMM patients treated with lenalidomide regimen: Newly diagnosed multiple myeloma patients who are not eligible for transplant and who are treated with a first-line regimen containing lenalidomide
  Interventions: Drug: Revlimid (lenalidomide)
- TNE NDMM patients treated with non-lenalidomide: Newly diagnosed multiple myeloma patients who are not eligible for transplant and who are treated with a first-line regimen not containing lenalidomide
  Interventions: Drug: Revlimid (lenalidomide)

INTERVENTIONS:
Drug: Revlimid (lenalidomide) — Treatment with first line Revlimid containing regimen as prescribed in routine clinical practice

SUMMARY:
This post authorization safety study is designed as prospective non interventional study for patients with newly diagnosed multiple myeloma who are not eligible for transplant. The objective is to compare the incidence of cardiovascular events between patients treated with a first-line lenalidomide containing regimen and those treated with a first-line non-lenalidomide containing regimen. Treatment in both cohorts will be done according to standard care. The study will gather risk factor information at baseline and throughout follow-up. Any cardiovascular event occurring will be assessed by an independent committee. Other safety endpoints will be collected through standard procedures. Observation period will be 3 years on treatment, with an additional evaluation of cardiovascular events 6 months' post treatment and a follow up period until 5 years after inclusion. During follow up the incidence of second primary malignancies (SPM) and overall survival will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Must have understood and voluntarily signed the Informed Consent Form (ICF)
2. Age ≥ 18 years at the time of signing the ICF
3. Newly diagnosed with multiple myeloma
4. Must not be eligible for transplant
5. Will be treated with a first-line lenalidomide-containing or nonlenalidomide-containing regimen, or currently is being treated with a first-line regimen and has received less than 2 cycles.

Exclusion Criteria:

1. Prior treatment for Monoclonal gammopathy of undetermined significance (MGUS) or smoldering myeloma with lenalidomide, thalidomide, or pomalidomide or any agent considered to be a first-line Multiple myeloma (MM) therapy.
2. Prior treatment with lenalidomide, thalidomide, or pomalidomide or any agent considered to be a first-line MM therapy through clinical trial participation or patient access program
3. Two or more complete cycles of first-line therapy or any agent considered to be a firstline MM therapy for newly diagnosed multiple myeloma (NDMM) treatment before study enrollment
4. Refusal to participate in the Revlimid Transplant noneligible (TNE) Newly diagnosed multiple myeloma (NDMM) Post-authorization safety study (PASS) or current participation in the treatment phase of an interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed multiple myeloma (NDMM) who are not eligible for transplant (TNE) starting their first treatment for multiple myeloma. Patients receiving any first line regimen can be included into the study. Decision for treatment needs to be done before inclusion into the trial.
Sampling Method: Non-Probability Sample
Enrollment: 911 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-01-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiovascular events | Approximately 8 years
  Number of participants with cardiovascular adverse events

SECONDARY OUTCOMES:
Incidence of renal impairment in NDMM patients | Approximately 8 years
  To document renal function among TNE NDMM patients treated with a first-line regimen
Incidence of infections in NDMM patients | Approximately 8 years
  To document the severity of infections among TNE NDMM patients treated with a first-line regimen.
Incidence of Second primary malignancy (SPM) in TNE NDMM patients treated with any first line regimen | Approximately 8 years
  Secondary primary malignancies will be categorized according to whether they are invasive and non-invasive malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, MD, Study Director — Bristol-Myers Squibb
Locations (125):
- Austria (3):
  - Innsbruck University Hospital, Innsbruck
  - LKH Hochsteiermark, Leoben
  - University hospital St. Pölten, Pölten
- Belgium (12):
  - CHU Saint-Pierre, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHU-Charleroi, Brussels
  - CHU-Charleroi, Charleroi
  - UZ Gent, Ghent
  - AZ Groeninge, Kortijk
  - CHR Citadelle Liège, Liège
  - Ziekehuis Oost Limburg, Limbourg
  - CHU Ambroise Pare, Mons
  - AZ Nikolaas, Sint Niklass
  - CHPLT Verviers, Verviers
  - CHU du Mont-Godinne, Yvoir
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Odense Hospital, Odense
- France (13):
  - Hôpital privé d'Antony - Ramsay Générale de Santé, Antony
  - CH Victor Dupouy, Argenteuil
  - Polyclinique Bordeaux Nord Aquaitaine, Bordeaux
  - Hospital Prive Sevigne, Cesson-Sévigné
  - GHM Institut Daniel Hollard, Grenoble
  - Clinique Victor Hugo, Le Mans
  - CH de Libourne, Libourne
  - CH Mont de Marsan, Mont-de-Marsan
  - CHU de Nice, Nice
  - CHR Orleans, Orléans
  - CH St Jean, Perpignan
  - Centre Hospitalier Universitaire (CHU) de Saint-Etienne - Hopital Nord, Saint-Etienne
  - Hospital Prive de Villeneuve d'Ascq, Villeneuve-d'Ascq
- Germany (30):
  - W8 Praxis für Onkologie, Aachen
  - Klinikum St. Marien Amberg, Amberg
  - Sozialstiftung Bamberg, Bamberg
  - Charité - Universitätsmedizin Berlin - Campus Charité Mitte, Berlin
  - Charité - Universitätsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Kliniken Berlin Köpenick, Berlin
  - HELIOS Klinikum Berlin Buch, Berlin
  - Gemeinschaftpraxis Pott/Tirier/Hannig, Bottrop
  - Onkologie Koln, Cologne
  - Medizinische Klinik II, DONAUISAR Klinikum Deggendorf, Akademisches Lehrkrankenhaus der Medizinischen Hochschule Hannover, Deggendorf
  - St. Bernward Krankenhaus GmbH, Hildesheim
  - Stadt. Krankenhaus Kiel, 2.med Klinik,, Kiel
  - Dres. Neise & Lollert, Praxis für Hämatologie & Onkologie, Krefeld
  - MVZ Mitte - Onkologische Schwerpunktpraxis, Leipzig
  - Lübecker Onkologische Schwerpunktpraxis, Lübeck
  - Klinikum Magdeburg, Magdeburg
  - Internistische Facharztzentrum mit Dialyse, Memmingen
  - Stauferklinikum, Mutlangen
  - Onko-Log Mulheim Gbr, Mülheim
  - Medizinisches Zentrum für Hämatologie und Onkologie München MVZ GmbH, München
  - Klinikum Nord, Klinik für Innere Medizin 5, Nuremberg
  - Onkologische Praxis Oldenburg, Oldenburg
  - Kreiskliniken Reutlingen, Reutlingen
  - Das Diak, Schwäbisch Hall
  - Klinikum Sindelfingen, Med.Klinik I, Sindelfingen
  - Onkologicum Stuttgart, Stuttgart
  - Ueboroertliche Berugsausuebungsgemeinschaft, Troisdorf
  - Kliniken Villingen-Schwenningen, Villingen-Schwenningen
  - Lahn-Dill-Kliniken, Wetzlar
  - Hämatologie / Internistische Onkologie, Wiesbaden
- Ireland (2):
  - Midlands Regional Hospital , Hematology/Oncology, Country Offaly
  - Waterford Regional Hospital, Waterford, Waterford
- Italy (30):
  - Ospedale di Ivrea, Chivasso, Corso Galileo Ferraris, 3 Chivasso
  - Ospedale Alessandria, Via Venezia, 16, 15121 Alessandria AL, Allessandria
  - Centro di Riferimento Oncologico di Aviano, Avianno
  - UO di Ematologia Osp. Mons Di Miccolis, Barletta
  - Istituto di Ematologia ed Ocnologia Medica "Seràgnoli" AUO Sant'Orsola - Bologna, Bologna
  - UO di Ematologia Osp. Perrino, Brindisi
  - Ospedale di Circolo di Busto Arsizio, Busto Arsizio
  - "S.C. di Ematologia e Centro Trapianti di Cellule Staminali Emopoietiche, Cagliari
  - Dipartimento di Oncologia Medica e Chirurgica AORN S. Anna e S. Sebastiano, Caserta
  - AO Garibaldi Catania - Via Palermo 636, Catania
  - AO Garibaldi Catania, Catania
  - Ospedale Ivrea , Areas Medica, Ivrea
  - Ospedale dell'Angelo, Mestre
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Opsedale di Bolzano, Milan
  - ASST Grande Ospedale Metropolitano Niguarda - Piazza Ospedale Maggiore, 3 -, Milan
  - Ospedale Maggiore di Novara, Novara
  - UO Ematologia e Centro Trapianti di Midollo Osseo dell'Ospedale San Francesco di Nuoro, Nuoro
  - IRCCS Policlinico di Pavia, Pavia
  - UO di Ematologia Osp. S. Carlo - Potenza, Potenza
  - Servizio immunoematologia e medicina trasfusionale-ASP, Ragusa
  - S.C. Ematologia, Dip.to Oncologico e Tecnologie Avanzate, Reggio Emilia
  - A.O Bianchi Melacrino Morelli - Presidio Riuniti, Regio Calabria
  - Ospedale Sant'Eugenio, Rome
  - Policlinico Gemelli Roma, Rome
  - UOSD Ematologia Complesso Opsedaliero-Ospedale S. Spirito e Nuovo Regina Margherita, Rome
  - Ospedale di Circolo, Fondazione Macchi, Varese
  - Ospdeale Policlinico Borgo Roma, Verona
  - Ospedale Belcolle Viterbo, Viterbo
- Netherlands (8):
  - Rode Kruis Hospital, Beverwijk
  - Nij Smellinghe, Drachten
  - Catharina Hospital, Hemato-Oncology, Eindhoven
  - Admiraal de Ruyter Hospital, Goes
  - Röpcke-Zweers Hospital, Hardenberg
  - Academic Hospital Maastricht, Maastricht
  - University Medical Center Utrecht, Utrecht
  - VieCuri Medical Center, Venlo
- Norway (2):
  - Helse Førde HF sentralsjukehuset, Førde
  - Akershus universitetssykehus HF, Lørenskog
- Spain (9):
  - Hospital de Jerez, Cadiz
  - Hospital Santa Lucía, Cartagena
  - Hospital de Jaen, Jaén
  - IP HULA, Lugo
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital Universitario Central Asturias, Oviedo
  - Son Espases, Palma de Mallorca
  - Complejo Universitario Navarra, Pamplona
  - Hospital Manises, Valencia
- Skåne University Hospital, Lund, Lund, Sweden
- United Kingdom (13):
  - Northern Health and Social Care Trust -Antrim Area Hospital, Antrim
  - South Eastern Health and Social Care Trust - The Ulster Hospital, Belfast
  - Birmingham Heartlands Hospital, Birmingham
  - Betsi Cadwaladr University Health Board - Glan Clwyd Hospital, Bodelwyddan
  - Southmead Hospital -North Bristol NHS Trust, Bristol
  - Queen Alexandra Hospital - Portsmouth Hospitals NHS Trust, Cosham
  - Lincoln County Hospital, Lincoln
  - The Clatterbridge Cancer Centre NHS Foundation Trust - The Royal Liverpool Hospital, Liverpool
  - St Georges Hospital, London
  - Norfolk and Norwich University Hospital, Norfolk
  - Southend Hospital, Southend-on-Sea
  - Royal Stoke Hospital, Stoke-on-Trent
  - Worcestershire Acute Hospitals NHS Trust - Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: No